CLINICAL TRIAL: NCT02041065
Title: Waterjet Versus Ultrasound Dissection During Hepatic Transection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Bengt Isaksson (Unknown); Jansson, Anders, M.D. (Individual)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011/2:4; 2011/2.4 (Other: Swedish Ethical Board)
Record Dates: First submitted 2013-10-09; First posted 2014-01-20 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Liver Tumour
Keywords: Liver transection; Bloodloss; Operation time; Safety; feasibility
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Waterjet induced dissection (Experimental): Waterjet induced dissection of the liver during resection.Waterjet dissection device mechanically separates hepatic tissue from bile ducts and vessels, the latter two to be separately ligated.
  Interventions: Device: Waterjet induced dissection
- CUSA induced dissection (Active Comparator): CUSA transection of the liver. Ultrasound based destruction of the liver parenchyma to allow separate ligation of the bile duct and intrahepatic vessels.
  Interventions: Device: CUSA induced dissection

INTERVENTIONS:
Device: Waterjet induced dissection — Waterjet induced dissection of the liver during resection.Waterjet dissection device mechanically separates hepatic tissue from bile ducts and vessels, the latter two to be separately ligated.
  Arms: Waterjet induced dissection
Device: CUSA induced dissection — Ultrasound based destruction of the liver
  Arms: CUSA induced dissection

SUMMARY:
Before liver transection patients are allocated to either waterjet or CUSA to divide the liver parenchyma.

DETAILED DESCRIPTION:
Transection time, bloodloss, total operation time and postoperative complication rates are registered.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic tumour suitable for resection
* patients 18 year or older Segmental resection Local resection Left sided hemihepatectomy

Exclusion Criteria:

* Right sided hemihepatectoyReresection In Situ Split Liver Extended left- and rightsided hemihepatectomy Lobus caudatus resection Central resections Hilus tumour/Klatskin/Cholangiocarcinoma Surgery on biliary tree Extended resection on other organs

Resection on gallbladder Resection on other organs during the same operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2011-02; Primary Completion 2015-02 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Peroperative bloodloss | During liver transection (on an average<90 min)
  Peroperative bloodloss in ml during liver transection by use of either waterjet or CUSA.

SECONDARY OUTCOMES:
Transection time in minutes | During liver transection (on an average< 90 minutes)
Operation time in minutes | Time spent in theater in minutes (on an average <240 minutes)
Hospital stay in days | Days spent in hospital after surgery (on an average < 10 days)

CONTACTS AND LOCATIONS:
Overall Officials: Anders Jansson, MdPhd, Study Chair — Karolinska University Hospital; Lars Lundell, Professor, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Centra of Gastroenterology, Stockholm, Sweden